CLINICAL TRIAL: NCT03874962
Title: Improvements in Pneumonia Status and Salivary Bacterial Concentration After Professional Oral Care Intervention in Taiwanese Nursing Home Residents
Brief Title: Improvements in Pneumonia Status After Oral Care Intervention in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KMUH103-3M47
Record Dates: First submitted 2018-04-18; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Pneumonia
Keywords: Oral care intervention; Nursing home residents
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine oral cleaning and professional oral care group (Experimental): The subjects in "Routine oral cleaning and professional oral care group" were received about routine oral cleaning and professional oral care.
  Interventions: Other: Routine oral cleaning and professional oral care group
- Routine oral cleaning group (No Intervention): The subjects in "Routine oral cleaning group" were received only routine oral cleaning, just maintain daily condition.

INTERVENTIONS:
Other: Routine oral cleaning and professional oral care group — Besides routine oral cleaning was conducted by caregivers, professional oral care intervention was conducted by dental hygienists, and it included muscle massage, oral cleaning, and oral health education once a week.
  Arms: Routine oral cleaning and professional oral care group

SUMMARY:
The correlation between improvement in oral health, reduction in oral bacterial concentration, and status of pneumonia hospitalization remains unclear. To determine the effects of professional oral care intervention on the index of oral health, salivary and sputum bacterial concentrations, and pneumonia hospitalization status of nursing home residents using a quasi-experimental study. Two nursing homes were on demand selected as the intervention and control groups; in the intervention group, weekly professional oral care was administered in addition to regular oral care by trained dental hygienists. Demographic data and oral health status were analyzed. Total salivary and sputum bacterial concentrations were determined using real-time polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* 51 year-old and above
* Being bedridden for ≥ 6 months
* Positive sputum production
* Difficulty in swallowing reported by caregivers

Exclusion Criteria:

* Below 51 year-old
* Patients or family refused any oral care

Ages: 51 Years to 102 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Pneumonia hospitalization status | 2 hours
  Hospitalization prevalence and days of each hospitalization due to pneumonia were collected from medical records by questionnaire.
Bacterial concentrations | 3 hours
  Total salivary and sputum bacterial concentrations were determined using real-time polymerase chain reaction. Staphylococcus aureus (strain ID: ATCC 29213) was used to create the standard growth curve of bacteria. After overnight culture, the samples were prepared by 5-fold serial dilution with normal saline and plating in a Petri dish to produce 2.5×103 to 3.9×107 CFU/mL of bacteria. Genomic DNA of bacteria was extracted from 1 mL of each bacterial serial solution using the modified standard method, which followed three basic steps: lysis, precipitation, and purification. The DNA extracts were resuspended in 20 µL of distilled water and stored at -80°C until real-time polymerase chain reaction (RT-PCR) amplification. The standard curve of bacterial concentration was generated by the bacterial 16S rRNA gene using a serial dilution of Staphylococcus aureus genomic DNA and StepOnePlus Real-Time PCR System (Applied Biosystems).

SECONDARY OUTCOMES:
Oral health examinations | 3 hours
  Oral health examinations were conducted by two trained dentists, and data on plaque, gingival, and tongue coating indexes were collected by oral examination tables.
Demographic data | 1 hour
  Demographic data included gender, age groups, conscious, educational level, and nutritional route, which were collected by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shun-Te Huang, Professor, Study Chair — Kaohsiung Medical University Chung-Ho Memorial Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD for outcome measures will be made available.
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication

REFERENCES:
- [Derived] Cao Y, Liu C, Lin J, Ng L, Needleman I, Walsh T, Li C. Oral care measures for preventing nursing home-acquired pneumonia. Cochrane Database Syst Rev. 2022 Nov 16;11(11):CD012416. doi: 10.1002/14651858.CD012416.pub3. PMID 36383760
- [Derived] Chiang TC, Huang MS, Lu PL, Huang ST, Lin YC. The effect of oral care intervention on pneumonia hospitalization, Staphylococcus aureus distribution, and salivary bacterial concentration in Taiwan nursing home residents: a pilot study. BMC Infect Dis. 2020 May 27;20(1):374. doi: 10.1186/s12879-020-05061-z. PMID 32460697